CLINICAL TRIAL: NCT06898203
Title: Precision Imaging to Evaluate Kaposi Sarcoma (PRIME-KS)
Brief Title: Precision Imaging to Evaluate Kaposi Sarcoma
Acronym: PRIME-KS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pensievision (Unknown); Kenya Medical Research Institute (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202411179; U01CA292765 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Kaposi Sarcoma
Keywords: Global Oncology; Kaposi Sarcoma; Affordable Cancer Technologies; Cancer in People with HIV; Human Centered Design; Discrete Choice Experiment; Medical devices; Low-cost design; Global health
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aim 2: Patients (Other): Patients will have three discrete skin lesions measured, with lesion area determined by ACTG criteria utilizing the product of longest perpendicular diameters. Patients will also have five 3D snapshots of each of the three target lesions taken, measuring lesion area automatically using SS3D.
  Interventions: Device: SkinScan3D
- Aim 3: Patients (Other): Providers will first measure KS lesions using the manual ruler-based method as per usual standard of care for the first three months. After the first three months, providers will switch to using SkinScan3D for KS skin lesion measurement.
  Interventions: Device: SkinScan3D

INTERVENTIONS:
Device: SkinScan3D — A handheld, simple, low-cost, and user-friendly technology that combines liquid lens technology and artificial intelligence (AI).
  Other Names: SS3D

SUMMARY:
AIM 1:

In Uganda and Kenya, Kaposi Sarcoma (KS) is one of the most common cancers and a leading cause of cancer-related deaths in men. However, tracking how well patients are responding to treatment is challenging, especially in busy clinics. Doctors must measure the size and changes in the areas affected by the cancer by hand, which can take a lot of time and can vary depending on the doctor. This method does not work well for patients with dark skin, which can lead to biases in treatment compared to patients with fairer skin.

To solve this problem, the investigators suggest the use of a simple, low-cost device that uses Artificial Intelligence (AI), the SkinScan3D (SS3D) device, to measure the cancer spots accurately and monitor changes over time. The goal of this study is to improve the SkinScan3D (SS3D) tool and the how it is used. The investigators will do this by talking to healthcare workers and patients, giving them surveys, and holding design workshops. The feedback from these activities will be shared with the device maker and local research teams to make the device better and ensure it is used properly.

AIMS 2 & 3:

In this study the investigators seek to formally compare reproducibility and accuracy of KS lesion size measurements between SkinScan3D and the current standard of care manual measurement method. The investigators will then test the SS3D device on 100 patients in a variety of real-world practice locations to determine whether the device will be usable, acceptable, appropriate, and feasible in routine care settings.

ELIGIBILITY:
Inclusion Criteria - Aim 2 (Patients):

* Adults age ≥18 years old
* Histopathology-confirmed Kaposi Sarcoma
* At least 3 skin lesions
* Capable of informed consent
* On treatment for Kaposi Sarcoma

Exclusion Criteria - Aim 2 (Patients):

* Patients not initiating Kaposi Sarcoma treatment
* Very ill patients requiring hospitalization

Inclusion Criteria - Aim 3 (Patients):

* Adults age ≥18 years old
* Histopathology-confirmed Kaposi Sarcoma
* Capable of informed consent
* Initiating treatment for Kaposi Sarcoma

Exclusion Criteria - Aim 3 (Patients):

* Patients with Kaposi Sarcoma that participated in Aim 1 or Aim 2
* Prior or ongoing Kaposi Sarcoma treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of KS lesion size measurements between SkinScan3D and current standard of care measurement - Aim 2 Only | Approximately 3 months
  Reproducibility/agreement between clinicians for each method is measured using the concordance correlation coefficient (CCC). A higher CCC means a more reproducible method.
Accuracy of KS lesion size measurements between SkinScan3D and current standard of care measurement - Aim 2 Only | Approximately 3 months
  Accuracy is measured using the coefficient of determination (R-squared). The R-squared tells us how much variation is due to varying lesion size as measured by either method versus how much variation is due to random error. When the variation due to random error is small, the R-squared value is closer to 1; when the variation due to random error is large, the R-squared value is farther from 1.
Device usability - Aim 3 Only | 6 months
  Device usability will be measured using the System Usability Scale. The SUS will result in a single composite score for each individual and the scores will be averaged to result in a single overall usability score.
Acceptability - Aim 3 Only | 6 months
  Acceptability of Intervention Measure (AIM), present participants with a set of 4 questions regarding their perception of an intervention's acceptability, typically on a 5-point Likert scale (completely disagree to completely agree), then calculate the average score across all items, with higher scores indicating greater perceived acceptability of the intervention.
Appropriateness - Aim 3 Only | 6 months
  Intervention Appropriateness Measure (IAM), will present a set of four questions to healthcare providers about how well SS3D works in their context. Each item is rated on a Likert scale, with higher scores indicating greater perceived appropriateness.
Feasibility - Aim 3 Only | 6 months
  FIM (Feasibility of Intervention Measure), will give the four-item questionnaire to healthcare providers asking them to rate how feasible they believe a specific intervention is on a Likert scale, usually ranging from "completely disagree" to "completely agree"; a higher score indicates greater perceived feasibility, with the average score across all items representing the overall feasibility rating of the intervention in that context.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Odeny, MBChB, MPH, PhD, Principal Investigator — Washington University School of Medicine
Locations (2):
- Kenya Medical Research Institute, Kisumu, Kenya
- Infectious Diseases Institute, Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
All participants will consent to the sharing of aggregate de-identified quantitative and qualitative data. Any potentially identifying variables will be stripped from the public-use data in compliance with Washington University IRB policies and human subject protections. Participants will have the option to consent to sharing their identifiable survey data for future research and scholarly use as part of a data donation agreement. These identifiable data will be made available as a separate, identifiable dataset in WURD. All deidentified study data that are not designated as restricted use will be made available as public use data to the research community via the WURD or QDR. Data that are determined to be potentially identifying though indirect or deductive disclosure are provided under restricted data contract to users who have a valid research need and meet conditions of use.
Supporting Information: Study Protocol, SAP
Time Frame: All data associated with study will be made available at the time of the first publication associated with the data. We anticipate that this will occur approximately 12 months following the completion of field work and within the award period. Study data deposited in WURD and QDR will be available to the public in perpetuity. Datasets related to methodological publications will be shared at publication.
Access Criteria: Contact Dr. Thomas Odeny

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu
- See also: Related Info — https://www.kemri.go.ke/
- See also: Related Info — https://idi.mak.ac.ug/